CLINICAL TRIAL: NCT00000224
Title: Alternate-Day Buprenorphine. Phase V
Brief Title: Alternate-Day Buprenorphine. Phase V - 6
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: University of Vermont (Other)
Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-06969-6; R01-06969-6
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-04

CONDITIONS: Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine

SUMMARY:
The purpose of this study is to evaluate buprenorphine blockade challenge.

ELIGIBILITY:
Please contact site for information.

Ages: 30 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1993-02

PRIMARY OUTCOMES:
Drug use
Opioid withdrawal
Subjective dose estimate
Drug effect characteristics: ARCI
Physiological changes in: pupil diameter
Physiological changes in: blood pressure
Physiological changes in: heart rate
Physiological changes in: respiration
Physiological changes in: bup plasma levels

CONTACTS AND LOCATIONS:
Overall Officials: Warren Bickel, Ph.D., Principal Investigator — University of Vermont
Locations (1):
- Treatment Research Center, Burlington, Vermont, United States

REFERENCES:
- [Background] Bickel, Amass, Badger (in preparation) A double-blind controlled trial of buprenorphine dosing every 72 hours in opioid dependenct humans. Bickel, Amass, Badger (in preparation) A double-blind controlled trial of buprenorphine dosing every 72 hours in opioid dependent humans.